CLINICAL TRIAL: NCT07276399
Title: A Phase 3, Randomized, Open-Label, Multicenter Study of Amivantamab in Addition to Carboplatin and Pembrolizumab, Compared to Standard of Care Platinum and Pembrolizumab and 5-FU, in Participants With Treatment-Naïve Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Amivantamab in Addition to Standard of Care Agents (SOC) Compared With SOC Alone in Participants With Recurrent/Metastatic Head and Neck Cancer
Acronym: OrigAMI-5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372HNC3001; 61186372HNC3001 (Other: Janssen Research & Development, LLC); 2025-521917-24-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — amivantamab; pembrolizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: Pembrolizumab, Amivantamab, Carboplatin (Experimental): Participants will receive pembrolizumab, amivantamab and carboplatin.
  Interventions: Biological: Amivantamab; Biological: Pembrolizumab; Drug: Carboplatin
- Arm B: Pembrolizumab, 5-Flurouracil (5-FU), Carboplatin or Cisplatin (Active Comparator): Participants will receive pembrolizumab, 5-FU and carboplatin or cisplatin (platinum therapy).
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: 5-Flurouracil; Drug: Cisplatin

INTERVENTIONS:
Biological: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372; RYBREVANT
  Arms: Arm A: Pembrolizumab, Amivantamab, Carboplatin
Biological: Pembrolizumab — Pembrolizumab will be administered.
Drug: Carboplatin — Carboplatin will be administered.
Drug: 5-Flurouracil — 5-Flurouracil will be administered for over 4-day infusion period.
  Arms: Arm B: Pembrolizumab, 5-Flurouracil (5-FU), Carboplatin or Cisplatin
Drug: Cisplatin — Cisplatin will be administered.
  Arms: Arm B: Pembrolizumab, 5-Flurouracil (5-FU), Carboplatin or Cisplatin

SUMMARY:
The purpose of this study is to compare anti-tumor activity of amivantamab in addition to pembrolizumab and carboplatin versus pembrolizumab, 5-fluorouracil (FU), and platinum therapy (carboplatin or cisplatin) in participants with refractory/metastatic (R/M) head and neck squamous cell carcinoma (HNSCC). HNSCC is a type of cancer that develops in the head and neck regions, including the outer tissue layer of the mouth and throat. This study will focus on participants with HNSCC who are treatment-naive (have not received prior treatment) in the R/M setting.

ELIGIBILITY:
Inclusion criteria:

* Be more than or equal to (>=) 18 years of age (or the legal age of majority in the jurisdiction in which the study is taking place, whichever is greater)
* Have histologically or cytologically confirmed recurrent/metastatic (R/M) HNSCC that is considered incurable by local therapies: a. eligible primary tumor locations are the oral cavity, oropharynx, hypopharynx, or larynx; b. Must not have a primary tumor site of nasopharynx or primary tumor of unknown location; c. Must have documented local testing results per local regulations; d. Human papillomavirus (HPV) status must be known for participants with primary tumor location in oropharynx via p16 test, HPV DNA test, or high-risk HPV in situ hybridization (ISH). Any known p16, HPV DNA, or high-risk HPV ISH status of tumor must be negative
* Be treatment-naive for systemic therapy in the R/M setting
* Have an ECOG performance status of 0 or 1
* Have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v).1.1

Exclusion criteria:

* Have an uncontrolled illness
* Have untreated brain metastases or history of known presence of leptomeningeal disease
* Have a history of clinically significant cardiovascular disease
* Inadequate organ or bone marrow function
* Known allergies, hypersensitivity, contraindications, or intolerance to excipients of: Amivantamab, Pembrolizumab, Carboplatin, Cisplatin, 5-FU and Hyaluronidase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-06-18 (Estimated); Study Completion 2029-06-18 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3 years 7 months
  OS is defined as time from the date of randomization to the date of death due to any cause.
Objective Response Rate (ORR) Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 3 years 7 months
  ORR is defined as the percentage of randomized participants achieving a confirmed best overall response (BOR) of partial response (PR) or complete response (CR) by BICR using RECIST version 1.1 .

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Using RECIST Version 1.1, as Assessed by BICR | Up to approximately 3 years 7 months
  PFS is defined as the time from randomization until the date of objective disease progression or death (due to any cause), whichever comes first, based on BICR assessment using RECIST v1.1, regardless of treatment discontinuation or start of subsequent anticancer therapy.
Duration of Response (DOR) As Assessed by BICR | Up to approximately 3 years 7 months
  DOR as assessed by BICR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR as best response.
ORR as Assessed by Investigator | Up to approximately 3 years 7 months
  ORR as assessed by the investigator is defined as the percentage of randomized participants achieving CR or PR, as defined by investigator assessment using RECIST v1.1 criteria.
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 3 years 7 months
  TEAE is defined as any new or worsening adverse event (AE) occurring at or after the initial administration of study treatment through the day of last dose plus 30 days or prior to the start of subsequent anticancer therapy, whichever is earlier, or any follow-up AE with onset date and time beyond 30 days after the last dose of study treatment but prior to the start of subsequent therapy or any AE that is considered treatment-related regardless of the start date of the event.
Number of Participants with Laboratory Abnormalities | Up to approximately 3 years 7 months
  Blood samples will be collected to determine the laboratory (serum chemistry and hematology) abnormalities.
Percentage of Participants with Improved or Stable Symptoms Compared to Baseline as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck Module 43 (EORTC QLQ-HN43) Symptom Scale Score | Baseline, up to approximately 3 years 7 months
  EORTC QLQ-HN43, is a self-administered, 43-item questionnaire measuring the health-related quality of life (HRQoL) of participants with head and neck cancer. EORTC QLQ-HN43 includes 19 scales (anxiety, body image, coughing, dry mouth and sticky saliva, neurological problems, opening mouth, pain in the mouth, social contact, problems with senses, shoulder problems, skin problems, swelling in the neck, social eating, speech, swallowing, sexuality, problems with teeth, weight loss, and problems with wound healing). Responses to items are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Higher scores indicate worse health outcomes.
Percentage of Participants with Improved or Stable Symptoms Compared to Baseline as Measured by EORTC QLQ-Core (C) 30 Symptom Scale Score | Baseline, up to approximately 3 years 7 months
  EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 3 symptom scales (fatigue, pain, and nausea and vomiting), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, or more severe symptoms.
Change from Baseline in Functioning HRQoL, as Measured by Functioning Scales of the EORTC QLQ-C30 | Baseline, up to approximately 3 years 7 months
  EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status / quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, or more severe symptoms.
Change from Baseline in Overall HRQoL, as Measured by Global Health Scales of the EORTC QLQ-C30 | Baseline, up to approximately 3 years 7 months
  EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the HRQoL of participants with cancer. EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status / quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, or more severe symptoms.
Differences Between Treatment Groups (Arms A and B) for EORTC Quality of Life (QLG) Item Library-46 (IL-46) Tolerability Scale Scores | Up to approximately 3 years 7 months
  EORTC IL46 is a single item used to measure the overall impact of treatment side effects. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Higher score indicates more impact of treatment side-effects.
Serum Concentration of Amivantamab | Up to approximately 3 years 7 months
  Serum concentrations of amivantamab will be analyzed.
Number of Participants with Serum Anti-Amivantamab Antibodies | Up to approximately 3 years 7 months
  Participants who are positive to serum anti-amivantamab antibodies will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (22):
- United States (11):
  - Providence St Jude Medical Center, Fullerton, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Central Georgia Cancer Care, Macon, Georgia
  - Cancer Care Specialists of Central Illinois, O'Fallon, Illinois
  - NHO Revive Research Institute, LLC, Lincoln, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Carolina Cancer Research Center, Wilson, North Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Arlington, Virginia
- St John of God Hospital Murdoch, Murdoch, Australia
- Brazil (4):
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto - Centro Integrado de Pesquisa, São José do Rio Preto
  - Associacao Feminina de Educacao e Combate ao Cancer Hospital Santa Rita de Cassia, Vitória
- Shanghai East Hospital, Shanghai, China
- Japan (3):
  - Hokkaido University Hospital, Sapporo
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City, Taiwan
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency